CLINICAL TRIAL: NCT01132963
Title: A Prospective Randomised Crossover Study to Evaluate the Effect Different Footwear Type Has on Measures of Balance and Confidence in Older Hospital Inpatients
Brief Title: The Effects of Footwear on Balance and Confidence in Older Inpatients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Dr Elizabeth Burleigh, NHS Greater Glasgow and Clyde
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: GN09GE487
Record Dates: First submitted 2010-05-27; First posted 2010-05-28 (Estimated); Last update posted 2010-05-28 (Estimated); Status verified 2010-03

CONDITIONS: Postural Balance; Accidental Falls

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Outdoor Shoes (Experimental): Patient will be asked to do balance tests while wearing outdoor shoes.
  Interventions: Other: Outdoor Shoes
- Pillow Paws Slippers (Active Comparator): Patient will be asked to complete balance tests while wearing standard hospital issue 'Pillow Paw' slippers on their feet
  Interventions: Other: Pillow Paw Slippers

INTERVENTIONS:
Other: Outdoor Shoes — Patient will be wearing sturdy outdoor shoes to complete balance tests
  Arms: Outdoor Shoes
Other: Pillow Paw Slippers — Patient will be wearing Pillow Paws slippers to complete balance tests which are issued to patients who do not have shoes in NHS hospitals in the UK
  Arms: Pillow Paws Slippers

SUMMARY:
The study aims to assess whether type of footwear worn changes the balance, mobility and confidence of older inpatients and consequently may affect their falls risk whilst in hospital. The investigators hope to identify which footwear type is most beneficial to patients in the ward environment.

DETAILED DESCRIPTION:
Footwear is known to be one of many recognised significant risk factors for falls, presumably by affecting balance and gait pattern. However, little is known regarding the best footwear for hospital inpatients in whom approximately 40% of older persons fall during their hospital admission. Patients admitted to hospital without their own footwear (slippers or shoes) are routinely given foam slippers referred to as pillow paws (PPs). There are concerns that these PPs may contribute to falls as they are often ill fitting (come in a very limited size range) and or are flimsy offering little foot and ankle support. Hence Medicine for the Elderly consultant and registrars designed this study to gain information on differences in balance, mobility and confidence when patients are wearing different footwear types. As a secondary outcome, falls data will also be collected to see whether there is any association between footwear types and inpatient falls incidence.

The aim is to compare pillow paws (PPs) with sturdy outdoor footwear or sturdy slippers. In this way we hope to gain information on which footwear type is most beneficial to hospital inpatients. A recent similar study infers that sturdy outdoor footwear benefits outpatients, but it is not clear whether the same applies to a hospital inpatient population whom are often frailer with greater co-morbidities (physical and mental) and a higher falls risk.

ELIGIBILITY:
Inclusion Criteria:

* Appropriate footwear
* Over 65 years
* Able to stand independently
* Inpatient in an acute geriatric assessment or rehabilitation ward

Exclusion Criteria:

* Unable to stand independently
* Acutely unwell
* Terminally unwell
* Registered partially sighted or blind
* Using lower limb orthotic device

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-11 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Functional Reach (centimeters) | Day 1 (at time of single assessment)
  Functional reach (FR):This is a measure of balance routinely performed on rehabilitation wards.
  The patient stands against a wall with one shoulder touching the wall and that arm fully extended horizontally. A mark is made on the wall recording the furthest point they are reaching to. They are then asked to stretch this arm as far forwards as they can without overbalancing/ stepping forwards. Another mark is made recording this maximum stretching distance. The difference between the 2 marks (in cm) is FR.
Timed Get-Up-And-Go (seconds) | Day 1 (at time of single assessment)
  Timed Get-Up-And-Go (TUG):- This is a measure of mobility that is recommended in guidelines for General Practitioners and hospital clinicians to perform as part of a simple falls risk assessment. The patient is timed on how long (IN SECONDS)it takes them to rise from a standard arm chair, walk to a line on the floor approx 10 feet away from chair, turn and return to the chair and sit back down.
The 4-point bedside balance score (0-4) | Day 1 (at time of single assessment)
  The 4-point bedside balance score:- This also assesses participants' balance. The patient's ability to stand with feet together, then with one foot slightly in front of the other (ie. standing partially heel to toe), followed by standing with one foot directly in front of the other (ie. standing fully heel to toe) and then standing on one leg is recorded. Increasing points are scored for each movement completed successfully. If it is clear that a patient cannot complete a particular movement, then the next level up in difficulty is not attempted.
Short Falls Efficiency Scale - International Questionnaire (score 7-28 points) | Day 1 (at time of single assessment)
  Short Falls Efficiency Scale - International (Short FES-I questionnaire) The patient will then be asked questions from the Short FES-I questionnaire. This asks the patient how concerned they would be about falling in the two footwear types in seven different situations. This is important to assess the influence footwear has on confidence.

SECONDARY OUTCOMES:
Incidence of falls during inpatient hospital stay | Variable - duration of hospital admission
  Any falls occurring during the participant's hospital stay will be recorded along with information on footwear worn at time of fall. This information can be accessed through NHS DATIX computerised incident reporting system.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Burleigh, MBChB MRCP, Study Director — NHS Greater Glasgow and Clyde; Alison Craig, MBChB MRCP, Principal Investigator — NHS Greater Glasgow and Clyde; Claire Steel, MBChB MRCP, Principal Investigator — NHS Greater Glasgow and Clyde; Jennifer Tilston, MBChB MRCP, Principal Investigator — NHS Greater Glasgow and Clyde; Lynsey Fielden, MBChB MRCP, Principal Investigator — NHS Greater Glasgow and Clyde; Steven Wishart, MBChB MRCP, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (4):
- United Kingdom (4):
  - Stobhill Hospital, Glasgow, Lanarkshire
  - Glasgow Royal Infirmary, Glasgow, Lanarkshire
  - Mansionhouse Unit, Victoria Infirmary, Glasgow, Lanarkshire
  - Southern General Hospital, Glasgow, Lanarkshire

REFERENCES:
- [Background] Menz HB, Lord SR. Footwear and postural stability in older people. J Am Podiatr Med Assoc. 1999 Jul;89(7):346-57. doi: 10.7547/87507315-89-7-346. PMID 10423940
- [Background] Horgan NF, Crehan F, Bartlett E, Keogan F, O'Grady AM, Moore AR, Donegan CF, Curran M. The effects of usual footwear on balance amongst elderly women attending a day hospital. Age Ageing. 2009 Jan;38(1):62-7. doi: 10.1093/ageing/afn219. Epub 2008 Nov 11. PMID 19001558
- [Background] Lord SR, Bashford GM. Shoe characteristics and balance in older women. J Am Geriatr Soc. 1996 Apr;44(4):429-33. doi: 10.1111/j.1532-5415.1996.tb06416.x. PMID 8636591
- [Background] Jessup RL. Foot pathology and inappropriate footwear as risk factors for falls in a subacute aged-care hospital. J Am Podiatr Med Assoc. 2007 May-Jun;97(3):213-7. doi: 10.7547/0970213. PMID 17507530
- [Background] Burns SL, Leese GP, McMurdo ME. Older people and ill fitting shoes. Postgrad Med J. 2002 Jun;78(920):344-6. doi: 10.1136/pmj.78.920.344. PMID 12151688
- [Background] Fortinsky RH, Iannuzzi-Sucich M, Baker DI, Gottschalk M, King MB, Brown CJ, Tinetti ME. Fall-risk assessment and management in clinical practice: views from healthcare providers. J Am Geriatr Soc. 2004 Sep;52(9):1522-6. doi: 10.1111/j.1532-5415.2004.52416.x. PMID 15341555
- [Background] Menant JC, Steele JR, Menz HB, Munro BJ, Lord SR. Effects of footwear features on balance and stepping in older people. Gerontology. 2008;54(1):18-23. doi: 10.1159/000115850. Epub 2008 Feb 4. PMID 18253023
- [Background] Tencer AF, Koepsell TD, Wolf ME, Frankenfeld CL, Buchner DM, Kukull WA, LaCroix AZ, Larson EB, Tautvydas M. Biomechanical properties of shoes and risk of falls in older adults. J Am Geriatr Soc. 2004 Nov;52(11):1840-6. doi: 10.1111/j.1532-5415.2004.52507.x. PMID 15507060
- [Background] Menz HB, Morris ME. Footwear characteristics and foot problems in older people. Gerontology. 2005 Sep-Oct;51(5):346-51. doi: 10.1159/000086373. PMID 16110238
- [Background] Koepsell TD, Wolf ME, Buchner DM, Kukull WA, LaCroix AZ, Tencer AF, Frankenfeld CL, Tautvydas M, Larson EB. Footwear style and risk of falls in older adults. J Am Geriatr Soc. 2004 Sep;52(9):1495-501. doi: 10.1111/j.1532-5415.2004.52412.x. PMID 15341551